CLINICAL TRIAL: NCT06983990
Title: Evaluation of the Relationship of Oxygen Reserve Index (ORI) and End-Tidal Carbon Dioxide (ETCO₂) With Arterial Blood Gas Parameters During the Apnea Test
Brief Title: ORI and ETCO₂ Relationship With Arterial Blood Gas During Apnea Test
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nilay Sertdemir, Resident Physician in Anesthesiology and Reanimation, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2023/05-06
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Brain Death
Keywords: Oxygen Reserve Index; ORI; Apnea test; Brain Death; End-Tidal Carbon Dioxide; ETCO2; Hyperoxia; Hypoxia
MeSH Terms: conditions — Brain Death; Hyperoxia; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apnea test group: Patients undergoing an apnea test as part of brain death evaluation are monitored for correlation analysis of oxygen reserve index (ORI), end-tidal CO₂ (ETCO₂), and arterial blood gas parameters (PaO₂, PaCO₂). No intervention is applied in this observational study.
  Interventions: Other: No intervention (observational monitoring only)

INTERVENTIONS:
Other: No intervention (observational monitoring only) — No intervention is applied. This is an observational study evaluating the correlation between non-invasive monitoring parameters and arterial blood gas values during apnea testing.

SUMMARY:
This observational study aims to evaluate the relationship between the Oxygen Reserve Index (ORI) and End-Tidal Carbon Dioxide (ETCO2) values with arterial blood gas parameters in patients undergoing the apnea test for the diagnosis of brain death. The study will examine the correlation between ORI and PaO2, as well as between ETCO2 and PaCO2. The primary objective is to assess the effectiveness of ORI in evaluating oxygenation and its applicability in the apnea test. The study will also evaluate the routine use of ORI in monitoring PaO2 and its potential benefits compared to traditional methods.

DETAILED DESCRIPTION:
This observational study aims to evaluate the relationship between the Oxygen Reserve Index (ORI) and partial arterial oxygen pressure (PaO2), as well as between End-Tidal Carbon Dioxide (ETCO2) and partial arterial carbon dioxide pressure (PaCO2) in patients undergoing an apnea test for the diagnosis of brain death. ORI is a relatively new, non-invasive monitoring tool that allows continuous and real-time assessment of oxygenation status. It is a dimensionless parameter with values ranging from 0 to 1. ORI is based on a multi-wavelength pulse co-oximeter that detects light absorption in both arterial and venous blood through a probe. It is designed to estimate PaO2 values in the 100-200 mmHg range, as SpO2 typically reaches ≥97% when PaO2 exceeds 80 mmHg, making it unable to reflect higher PaO2 levels accurately. The apnea test is a critical procedure for the diagnosis of brain death, in which the presence or absence of spontaneous breathing in response to carbon dioxide accumulation is evaluated. During the test, arterial blood gas (ABG) measurements are taken to monitor the rise in PaCO2. Before the test begins, the patient is ventilated with 100% oxygen to raise PaO2 above 200 mmHg, which is confirmed with a pre-test ABG sample. The patient must also be normocapnic prior to testing.

As arterial blood sampling is an invasive procedure, this study aims to assess the predictability of PaO2 and PaCO2 using ORI and ETCO2 in the pre-test phase. The primary objective is to determine the capability of ORI to monitor oxygenation status and evaluate its potential to detect hypoxia earlier. Moreover, by comparing ORI to conventional methods, this study seeks to explore its potential routine use in clinical settings for PaO2 monitoring and its possible advantages. In patients undergoing apnea testing for suspected brain death, this study may help determine whether ORI offers benefits over current monitoring approaches and whether it can reduce dependence on invasive ABG sampling. Furthermore, hyperoxia, like hypoxia, poses various clinical risks. The clinical use of ORI alongside SpO2 may help prevent hyperoxia and enable earlier detection of hypoxia. This may enhance patient safety and improve clinical decision-making in critical care environments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all the prerequisites for initiating the brain death diagnosis process and for whom the decision to perform the apnea test for diagnosis of brain death.
* Patients aged 18 years or older.
* Patients who have provided verbal and written consent from their first-degree relatives.

Exclusion Criteria:

* Patients whose first-degree relatives do not consent to participation in the study.
* Patients in whom the ORI probe cannot be used due to circulatory disturbances in the extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients (aged 18 and over) who are being monitored in the intensive care units of the University of Health Sciences Bursa Yuksek Ihtisas Training and Research Hospital and are suspected of brain death, for whom an apnea test has been scheduled by their physician as part of the brain death diagnosis process. The study population will consist of patients who meet the inclusion criteria and for whom written informed consent has been obtained from a legally authorized representative. Patients whose first-degree relatives have declined participation, and those in whom the Oxygen Reserve Index (ORI) probe cannot be used due to circulatory disorders in the extremities, will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between Oxygen Reserve Index (ORI) and arterial PaO2 during apnea test | Before and at specific intervals during the apnea test
  Assess the correlation between non-invasive ORI values obtained from Masimo pulse CO-oximeter and arterial partial pressure of oxygen (PaO2) measured from arterial blood gases during the apnea test.

SECONDARY OUTCOMES:
Correlation between End-Tidal Carbon Dioxide (ETCO2) and arterial PaCO2 during apnea test | Before the apnea test, at the start of the test, and end of the test
  Assess the correlation between ETCO2 values from capnography and arterial partial pressure of carbon dioxide (PaCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Nilay SERTDEMIR, MD, Principal Investigator — Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital
Locations (1):
- Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vivien B, Amour J, Nicolas-Robin A, Vesque M, Langeron O, Coriat P, Riou B. An evaluation of capnography monitoring during the apnoea test in brain-dead patients. Eur J Anaesthesiol. 2007 Oct;24(10):868-75. doi: 10.1017/S0265021507000725. Epub 2007 Jun 20. PMID 17579950
- [Background] Applegate RL 2nd, Dorotta IL, Wells B, Juma D, Applegate PM. The Relationship Between Oxygen Reserve Index and Arterial Partial Pressure of Oxygen During Surgery. Anesth Analg. 2016 Sep;123(3):626-33. doi: 10.1213/ANE.0000000000001262. PMID 27007078